CLINICAL TRIAL: NCT02366793
Title: Accessory Joint and Neural Mobilizations in Shoulder Range of Motion Restriction After Breast Cancer Surgery. A Pilot Randomized Clinical Trial.
Brief Title: Accessory Joint and Neural Mobilizations in Shoulder After Breast Cancer Surgery. Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, IRENE DE LA ROSA DÍAZ, Irene de la Rosa Díaz, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAlcala
Record Dates: First submitted 2015-01-17; First posted 2015-02-19 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: accessory mobilization, nerve mobilization.
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accessory joint mobilization (Experimental): Humeral head slides, anterior, posterior and caudal slides.
  Interventions: Other: Accessory joint mobilization
- Nerve mobilization (Experimental): neural tissue longitudinal slide using the median neurodynamic test 1 (Butler).
  Interventions: Other: Nerve mobilization

INTERVENTIONS:
Other: Accessory joint mobilization — Three kinds of humeral head slides: anterior, posterior and caudal slides. Subjects remained in supine position during the whole treatment. The techniques were applied in a rhythmical way, with 2 seconds of slide/traction and then a 2-second break. Each technique was carried out for 2 minutes.
  Arms: Accessory joint mobilization
Other: Nerve mobilization — Neural tissue longitudinal slide using the median neurodynamic test 1 (MNT1) that was described by Butler. The proximal parameters (scapular depression, abduction and humeral external rotation) were introduced with maximum neural tension. On the other hand, the distal parameters (supination, elbow extension, wrist and fingers extension) received the remaining tension that the neural tissue allowed. The parameters were introduced sequentially in the order exposed
  Arms: Nerve mobilization

SUMMARY:
The potential consequences after breast cancer surgery are joint pain and sensitive disorders, the main sign of which is alterations in shoulder mobility. Global kinesitherapy has been shown to be effective at increasing shoulder range of motion restriction. However, literature does not consider specific manual therapy techniques, which means peripheral nerves and articular capsule have not been taken into account. These two tissues are potentially damaged structures during surgery and they are main responsible for shoulder range of motion restriction The main objective of this study is to pilot the effectiveness of accessory joint and nerve mobilization techniques in order to get an overview of the articular capsule and nerve dysfunctions involvement in shoulder motion restriction.

DETAILED DESCRIPTION:
Background: The potential consequences after breast cancer surgery are joint pain and sensitive disorders, the main sign of which is alterations in shoulder mobility. Design: Prospective randomized and double-blind pilot trial. Objective: To pilot the effectiveness of accessory joint and nerve mobilization techniques in order to get an overview of the joint capsule and nerve involvement in shoulder motion restriction. Participants: 18 women who were undergoing unilateral breast cancer surgery and axillary lymph node dissection. Setting: Women´s Health Research Group at Physical Therapy Department of University of Alcala, Madrid, Spain. Intervention: accessory joint mobilization versus neural mobilization. Follow-up: Six-month follow-up. Key outcomes: Range of motion, sensitive disorder, pain and upper limb functionality.

ELIGIBILITY:
Inclusion Criteria:

* unilateral breast cancer diagnosis
* breast cancer with axillary lymph node dissection
* be willing to sign the informed consent form

Exclusion Criteria:

* bilateral breast cancer diagnosis
* loco-regional recurrence
* systemic disease
* had not undergone the axillary lymph node dissection approach
* to present any contraindication for Physical Therapy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Shoulder Range of motion | 15 min
  Shoulder movements measured: flexion, extension, abduction, external e internal rotation.
  Measure instrument: inclinometer. Unit of measure: degrees. Number of participants: 18.

SECONDARY OUTCOMES:
Pain | 5 min
  Measure instrument: Visual Analogue Scale to measure the grade of pain: scale from 0 (no pain) to 10 (unbearable pain). Patients choose where is located their pain throughout this scale.
  Unit of measure: from 0 to 10 points. Number of participants: 18.
Upper limb functionality | 10 min
  Measured items: daily life activities related to the upper limb such as to comb, to get washed, to button the bra, to mop the floor, to clean windows, to hang up, to make the bed, to carry the shopping cart, to put on the pullover, to take off the pullover, leisure.
  Measure instrument: the Wingate's Daily Life Activities Table to measure the daily life activities difficulty. Patients give a score of how difficult is each daily life activity. Score from 0 (no difficulty) to 3 (disability).
  Unit of measure: from 0 to 3 points. Number of participants: 18.

CONTACTS AND LOCATIONS:
Overall Officials: MARÍA TORRES-LACOMBA, DOCTOR, Study Director — SUPERVISOR